CLINICAL TRIAL: NCT00222768
Title: Three-Tracer PET Quantitation of Insulin Action in Muscle
Brief Title: PET Imaging of Regional Variation in Insulin Sensitivity of Adipose Tissue in Humans
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: 0502008; R01DK060555 (NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2008-02

CONDITIONS: Diabetes; Obesity
Keywords: Adipose tissue; PET imaging
MeSH Terms: conditions — Diabetes Mellitus; Obesity

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this research study is to use a relatively new technology, called Positron Emission Tomography (PET), to study how insulin works on sugar in your body's fatty tissue. PET imaging is a way of obtaining a "metabolic image" of your internal organs. It does not involve surgery and is not a high risk process. It has been used successfully to study brain, heart and more recently, skeletal muscle. In this research study, we will use PET in combination with Magnetic Resonance Imaging (MRI), to study fatty tissues in healthy people who do not have diabetes. In the future, we plan to do similar PET/MRI studies in individuals with type 2 diabetes mellitus (T2DM) and in individuals who are likely to develop T2DM.

Fat tissue might have a lot to do with developing type 2 diabetes. First, it is well recognized that excess fatty tissues, especially the kind in your belly, increases risk for the development of T2DM, as well as affecting other ways the body uses insulin. Second, fatty tissue is a classic target tissue for the action of insulin, which regulates the use of sugar by fat cells and also regulates the release of fatty acids from fatty tissues. Third, studies in mice that lack fatty tissue, indicate that severe insulin resistance (lack of a normal response to insulin) can result. Other types of studies have shown that fatty tissues make proteins that affect your body's insulin and your appetite in good and bad ways. Yet despite this importance, we still lack techniques for the study of fatty tissue metabolism in humans.

DETAILED DESCRIPTION:
The association of adiposity with insulin resistance (IR) is modulated by regional fat deposition. For example, visceral (intra-abdominal) adipose tissue (VAT) is generally regarded as more strongly correlated with IR, than subcutaneous adiposity of the thigh (ThiSAT) or abdomen (AbdSAT), even though these latter depots are larger than VAT. Perhaps these differences are due to regional variation in AT metabolism. A limitation of body composition methods is that these assess amount rather than metabolism of adipose tissue (AT). Our aim is to use positron emission tomography (PET) imaging with [F-18] fluorodeoxyglucose (FDG) for the in vivo investigation of AT metabolism and use this in conjunction with regional body composition imaging so that both the amount of AT and metabolism of AT can be determined. Hopefully, such an approach will give new insight as to how AT influences skeletal muscle and hepatic IR. The current project seeks to develop this approach, generating preliminary data to lay a foundation for subsequent projects.

The first specific aim is conduct dose-responsive measurement of insulin-stimulated glucose uptake (i.e. insulin sensitivity) of AT in humans using PET imaging in healthy volunteers. We will examine the effects of insulin infusion rates at 0, 20, and 80 mU/min-m2 body surface area.

The second specific aim is to assess regional variation in insulin-stimulated glucose uptake in AT, comparing VAT, AbdSAT and ThiSAT in volunteers without IR. We will test the hypothesis that insulin sensitivity (IS) follows the rank order of ThiSAT IS > AbdSAT IS > VAT IS.

At any given body mass index, fat mass constitutes a higher percentage of body weight in women than men. The third specific aim is to assess potential gender-differences in AT metabolism, testing the hypothesis that AT IS is greater in women than men.

ELIGIBILITY:
Inclusion Criteria:

* A thorough medical examination will be done at the screening examination. To be eligible for these studies, volunteers must be free of clinical evidence of cardiac, renal, hepatic, and vascular disease, or other major medical problems that would endanger the volunteers or compromise the scientific validity of the studies.

We will recruit 20 volunteers (10 men and 10 women), non-obese (BMI 20 to 27 kg/m2), glucose tolerant, healthy volunteers, who are between the ages of 25 and 45 years old. Volunteers for this study must have a fasting glucose < 100 mg/dl; HbA1c < 5.7%; Hct > 34; fasting plasma insulin level < 12 µU/ml; ALT < 60; AST < 60; Alk phos < 150; TSH < 6; Trig < 150 mg/dl; Chol < 250; systolic BP < 140; diastolic BP < 90; negative family history (first-degree relatives) for type 2 DM; be in good health and not be taking any chronic medications known to affect adipose tissue metabolism or insulin sensitivity (e.g. glucocorticoids, thiazide diuretics).

Exclusion Criteria:

* Pregnant women and women who are currently breast-feeding will be excluded from study participation. Women will be checked for pregnancy (using a urine pregnancy test) at screening, within 24 hours prior to the DEXA scan and within 24 hours prior to each PET and MRI study. Previous difficulty with xylocaine or claustrophobia will exclude.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20
Dates: Start 2005-04; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Method development of dose-responsive measurement of insulin-stimulated glucose uptake of adipose tissue using 18-FDG and Positron Emission Tomography

SECONDARY OUTCOMES:
To assess regional variation in insulin-stimulated glucose uptake in adipose tissue.

CONTACTS AND LOCATIONS:
Overall Officials: David E. Kelley, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States